CLINICAL TRIAL: NCT04480606
Title: Effects of Home Exercise Program Applied to the Socially Isolated Elderly Due to COVID-19 on Physical Activity Level, Functional Capacity and Quality of Life
Brief Title: Evaluation of the Physical Activity Level of the Elderly in Social Isolation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 008
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Exercise Program
Keywords: elderly; COVID 19; physical activity
MeSH Terms: conditions — COVID-19; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home exercise group (Experimental): 47 volunteers over 65 years old who are at home during the social isolation process due to the coronavirus outbreak will be included in home exercise group.
  Interventions: Behavioral: Home exercise program
- Control Group (No Intervention): The control group will be asked to remain isolated as they are and the exercise program will not be implemented.

INTERVENTIONS:
Behavioral: Home exercise program — 47 volunteers over 65 years old who are at home during the social isolation process due to the coronavirus outbreak will be included in home exercise group. A video exercise protocol was created and each exercise session was planned as daily 30 minutes for 6 weeks. Individuals will ask to do their exercises. It was planned to start the protocol with warm-up exercises and finish with cooling exercises. The exercise protocol was additionally determined as a combination of aerobic, balance and strengthening exercises. The exercise program consists of 3 levels and individuals will be provided to start at a level appropriate to their level of physical activity.
  Arms: Home exercise group

SUMMARY:
Due to the COVID-19 pandemic in our country, individuals over 65 are prohibited from leaving their homes by T.C. The Ministry of Internal Affairs on March 21, 2020. While social isolation provides protection from COVID-19, it also brings some side effects that pose health risks. Studies investigating the relationship between social isolation and health behavior report that individuals with smaller social networks report less healthy diets, excessive alcohol consumption, and less physical activity. The effects of social isolation are related to physical inactivity, smoking.

Physical activity is any body movement produced by the contraction of skeletal muscles that increases energy consumption. 150 minutes of moderate PA, 75 minutes of severe PA per week, or combined moderate and severe intensity PA plus twice a week strength training is recommended for elderly. The prevalence of physical inactivity increases significantly with increasing age. At the global level, approximately 45% of people over the age of 60 do not meet the recommended level of PA. The decrease in physical performance is associated with the risk of falling, sarcopenia, fragility, decreased quality of life, emotionalization, comorbidity, early death, and increased health care costs.

The purpose of this study; to evaluate the physical activity level, functional capacity and quality of life of individuals over the age of 65 who socially isolated due to the precautions COVID-19 pandemic, and to investigate the effectiveness of video based home exercise program.

DETAILED DESCRIPTION:
94 volunteers over 65 years old who are at home during the social isolation process due to the coronavirus outbreak will be included in the study. Participants will be divided into 2 groups of 47 people. 47 volunteers over 65 years old who are at home during the social isolation process due to the coronavirus outbreak will be included in home exercise group. A video exercise protocol was created and each exercise session was planned as daily 30 minutes for 6 weeks. Individuals will ask to do their exercises. It was planned to start the protocol with warm-up exercises and finish with cooling exercises. The exercise protocol was additionally determined as a combination of aerobic, balance and strengthening exercises. The exercise program consists of 3 levels and individuals will be provided to start at a level appropriate to their level of physical activity. The control group will be asked to remain isolated as they are and the exercise program will not be implemented.

Evaluation methods will be applied before starting the exercise program and at the end of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years old and over
* Being in social isolation due to coronavirus epidemic
* Spending at least 1 week at home different from routine life
* Not to be obstructed from doing physical activities
* To have access to online exercise training

Exclusion Criteria:

* Having serious cognitive impairment (Mini-mental state examination being lower than 24)
* Having serious hearing and vision problems
* Having vestibular disorders that can cause loss of balance
* having serious heart disease (aortic stenosis, angina, hypertrophic cardiac myopathy, arrhythmia, pacemaker)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-11-20 (Estimated); Study Completion 2020-11-20 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Scale for the Elderly | 6 weeks
  Physical Activity Scale for the Elderly will use to assess the physical activity level of elderly individuals, the factors affecting the activity level, the relationship between physical activity and health profile. The minimum and maximum score that can be obtained from the scale is 0 and 400.The higher score indicates better level of physical activity.
Nottingham Health Profile | 6 weeks
  Nottingham Health Profile will use to assess the quality of life related to health. It is a general quality of life questionnaire that assesses the level of individuals' health problems and how they affect their daily life activities. It have six subtitles, scored between 0-100. The high total score indicates that the health condition is bad.
Short Physical Performance Battery | 6 weeks
  Short Physical Performance Battery will use to assess physical performance. This test consists of 3 objective tests that evaluate lower body function; 4 meters walking, getting up from the chair and standing balance test. 5-step (0-4) summary score is assigned for each test; higher scores show better physical performance.

SECONDARY OUTCOMES:
Beck anxiety inventory | 6 weeks
  Beck anxiety inventory will use to assess anxiety level. The survey includes substances that determine anxious temperament, autonomic hyperactivity and motor tension, some cognitions. The patient is asked to evaluate the symptoms within the 'last week including today'. Each symptom is evaluated as none, mild, moderate, and severe. The total score ranges from 0-63.
Beck depression inventory | 6 weeks
  Beck depression inventory will use to assess depression level. It consists of 21 items with an increasing score between 0-3. The total score ranges from 0-63.
Contentment With Life Scale | 6 weeks
  Contentment With Life Scale will use to assess satisfaction level. The questionnaire consists of 5 questions in total and each question has a threshold of evaluation from 5 to 25 points (5 points for the worst and 25 points for the best).

IPD SHARING:
Plan to Share IPD: No